CLINICAL TRIAL: NCT02843230
Title: Monitoring Anti-angiogenic Therapy in Brain Tumors by Advanced MRI
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Eva Maria Ratai, PhD, Massachusetts General Hospital
Other Study IDs: 16-147
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Glioblastoma
Keywords: Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Bevacizumab; Lomustine; Temozolomide; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Avastin Combine with MRI, DSC and MRS Scan: Study subjects will have an MRI exam including MRS and DSC imaging prior to bevacizumab/ Avastin treatment (baseline scan).
  * Subsequently, patients will receive their follow-up MRI exams every 8 weeks as standard of care.
  * Advanced imaging will be added to the patients' regular follow-up scans including MRS and DSC MRI.
  Interventions: Radiation: Avastin; Device: MRI; Device: MRS; Device: DSC
- Avastin and Temozolomide Combine with DSC, MRI and MRS Scan: Study subjects will have an MRI exam including MRS and DSC imaging prior to bevacizumab/ Avastin and Temozolomide treatment (baseline scan).
  * Subsequently, patients will receive their follow-up MRI exams every 8 weeks as standard of care.
  * Advanced imaging will be added to the patients' regular follow-up scans including MRS and DSC MRI.
  Interventions: Radiation: Avastin; Radiation: Temozolomide; Device: MRI; Device: MRS; Device: DSC
- Avastin and Lomustine Combine with MRI, DSC, and MRS Scan: Study subjects will have an MRI exam including MRS and DSC imaging prior to bevacizumab/ Avastin and Lomustine treatment (baseline scan).
  * Subsequently, patients will receive their follow-up MRI exams every 6 weeks as standard of care.
  * Advanced imaging will be added to the patients' regular follow-up scans including MRS and DSC MRI.
  Interventions: Radiation: Avastin; Radiation: Lomustine; Device: MRI; Device: MRS; Device: DSC

INTERVENTIONS:
Radiation: Avastin
  Other Names: Bevacizumab
Radiation: Lomustine
  Other Names: Ceenu
  Groups: Avastin and Lomustine Combine with MRI, DSC, and MRS Scan
Radiation: Temozolomide
  Other Names: Temodar
  Groups: Avastin and Temozolomide Combine with DSC, MRI and MRS Scan
Device: MRI
  Other Names: Magnetic Resonance Imaging
Device: MRS
  Other Names: Magnetic Resonance Spectroscopy
Device: DSC
  Other Names: Dynamic Susceptibility Contrast Imaging

SUMMARY:
This research study aims to predict treatment response to anti-angiogenic therapy (Avastin) using advanced magnetic resonance imaging (MRI) and spectroscopy (MRS) for Glioblastoma patients.

DETAILED DESCRIPTION:
This research study is an Imaging Study, in which investigators are examining if advanced magnetic resonance imaging (MRI) and spectroscopy (MRS) are able to predict the outcome of participants with a brain tumor (glioblastoma) treated with an anti-angiogenic treatment called Avastin (Avastin is the trade name for bevacizumab).

MRI studies the tumor size and other physical aspects of a tumor and the MRS adds an additional analysis that measures the chemical changes that a tumor undergoes. This study aims to test whether addition of MRS to standard MRI testing will help better predict how a tumor is responding to therapy.

The names of the study interventions involved in this study are:

* MRI/MRS
* Avastin Avastin works by interfering with the process of new blood vessel growth and is thus an anti-angiogenic. Avastin is approved by the U.S. Food and Drug Administration for use in Glioblastoma .

The participant's treating physician may complement the Avastin treatment with chemotherapy including Temozolomide (TMZ) or Lomustine (CCNU). Both treatments are approved by the U.S. Food and Drug Administration for use in Glioblastoma.

The purpose of this study is to predict treatment response to anti-angiogenic therapy in brain tumor participant using advanced MRI and MRS.

MRI/MRS is an FDA-approved test that uses magnets to take pictures of the brain and lets us "see inside" the body/brain without surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed glioblastoma and evidence of recurrence. Patients with low-grade tumors who have progressed to glioblastoma are eligible.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm.
* Patients must be anti-angiogenic therapy naïve.
* Age ≥18 years. We exclude children because the chances of recruiting children with recurrent glioblastoma who will be treated with bevacizumab are small.
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Life expectancy of greater than 10 weeks.

  * creatinine within normal institutional limits OR
  * creatinine clearance ≥30 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Participants must be able to undergo MRI scan.
* Participants whose clinical care plan includes treatment with bevacizumab mono-therapy (Group I) or bevacizumab (+ cytotoxic agents Temozolomide (TMZ) or Lomustine (CCNU).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have already received anti-VEGF or investigational anti-angiogenic therapy for glioblastoma.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the effects of MR imaging on the fetus are unknown and gadolinium-based intravenous contrast material is not recommended for use in pregnant patients
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with bevacizumab, Temozolomide (TMZ) or Lomustine (CCNU).
* Patients who are no suitable to undergo MRI or use gadolinium contrast due to:

  * Claustrophobia
  * Presence of metallic objects or implanted medical devices in body (i.e. cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
  * Sickle cell disease
  * Renal failure
  * Reduced renal function, as determined by creatinine clearance < 30 mL/min based on a serum creatinine level obtained within 28 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent glioblstoma
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival For Patients Receiving Advanced MRI and MRS | 6 months
Overall Survival For Patients Receiving Advanced MRI and MRS | 12 months

SECONDARY OUTCOMES:
Progression Free Survival For Patient Receiving Dynamic Susceptibility Contrast | 6 months
Overall Survival Rate For Patient Receiving Dynamic Susceptibility Contrast | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Eva-Maria Ratai, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Abtah ME, Wenke MR, Talati P, Fu M, Kim D, Weerasekera A, He J, Vaynrub A, Vangel M, Rapalino O, Andronesi O, Arrillaga-Romany I, Forst DA, Yen YF, Rosen B, Batchelor TT, Gonzalez RG, Dietrich J, Gerstner ER, Ratai EM. Myo-Inositol Levels Measured with MR Spectroscopy Can Help Predict Failure of Antiangiogenic Treatment in Recurrent Glioblastoma. Radiology. 2022 Feb;302(2):410-418. doi: 10.1148/radiol.2021210826. Epub 2021 Nov 9. PMID 34751617